CLINICAL TRIAL: NCT00006444
Title: Assessment of Prevalence and Persistence of Human Papillomavirus (HPV) DNA in HIV-Infected Women Who Are Antiretroviral Naive and Have Initiated HAART
Brief Title: The Effects of Combination Anti-HIV Medication on Human Papillomavirus (HPV) in HIV-Infected Women
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Other Study IDs: A5029; AACTG A5029; ACTG A5029
Record Dates: First submitted 2000-11-03; First posted 2001-08-31 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-11

CONDITIONS: HIV Infections; Papilloma
Keywords: Drug Therapy, Combination; Papillomavirus, Human; DNA, Viral; Anti-HIV Agent; Treatment Naive
MeSH Terms: conditions — HIV Infections; Papilloma

SUMMARY:
The purpose of this study is to see how often human papillomavirus (HPV) occurs in HIV-infected women who have not taken anti-HIV drugs and to learn whether taking anti-HIV drugs will affect HPV in women.

HIV infection increases the risk of getting HPV infection. Findings suggest that HIV infection as well as a weakened immune system may increase the chances of getting HPV. Aggressive anti-HIV medication has been shown to strengthen the immune system. Researchers want to learn whether anti-HIV drugs affect the HPV virus or decrease the chances of getting HPV. This study is important because it may provide important information to help manage a woman's health and to determine a woman's risk for developing problems with the cervix (outer end of the uterus).

DETAILED DESCRIPTION:
HIV infection is a significant risk factor for human HPV infection and the development of HPV-associated lesions in the female genital tract. Findings suggest that HIV infection and/or HIV-related immunosuppression increases a woman's susceptibility to HPV infection or alters the natural history of preexisting HPV infection. Treatment with HAART has been shown to result in significant increases in CD4+ cell counts and "partial reconstitution" of the immune system. It is not known whether treatment of HIV infection with potent antiretroviral regimens could affect the persistence of HPV infection and progression of cervical dysplasia. This study is important for HIV-infected women because of the implications for gynecologic management and determination of cervical disease risk.

At baseline, Weeks 24 and 48, and then every 48 weeks until study completion, women undergo pelvic examination and cervical specimens collection by the following methods: 1) Sno-strip; 2) cervicovaginal lavage; 3) cervical brush method; and 4) Pap smear. A colposcopy is required for any woman who has an abnormal Pap smear reading unless the abnormal Pap smear is thought to be due to an intercurrent infection. A cervical biopsy is strongly recommended in the event of an abnormal colposcopy. Blood is collected for HPV antibody testing, viral load, and CD4 measures.

ELIGIBILITY:
Inclusion Criteria

Women may be eligible for this study if they:

* Are HIV-positive.
* Are at least 13 years of age and menstruating.
* Are willing to enroll in another drug study.
* Have written consent of a parent or guardian if under 18 years.
* This study has been changed to increase enrollment. Women who are starting HAART-based therapy prescribed by a personal physician or participating in an antiretroviral trial are all eligible.
* Intend to start antiretroviral therapy within 14 days of study entry.

Exclusion Criteria

Women will not be eligible for this study if they:

* Have been on anti-HIV treatment for more than 14 days.
* Are abusing drugs or alcohol.
* Are receiving medication that affects the immune system, fights HPV, or is investigational, except for anti-HIV drugs provided by coenrolling in a Phase II or III trial with approval of a study chair within 30 days of study entry, including but not limited to systemic interferons and interleukins, thalidomide, systemic cidofovir, and HPV vaccines. This study has been changed. The following medications are no longer excluded: thymopentin, hydroxyurea, granulocyte colony-stimulating factor (G-CSF and filgrastim), and GM-CSF (sargramostim).
* Have cervical cancer or a history of cervical cancer.
* Have had a hysterectomy (removal of the uterus).
* Participated in HPV trials at any time.
* Use imiquimod inside the vagina.
* Are taking corticosteroid treatment in large doses.

Min Age: 13 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160
Dates: Start 2000-11; Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Squires, Study Chair; Rebecca Clark, Study Chair; Kenneth H Fife, Study Chair
Locations (51):
- United States (49):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - Children's Hosp of Los Angeles/UCLA Med Ctr, Los Angeles, California
  - Univ of Southern California / LA County USC Med Ctr, Los Angeles, California
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - UCLA CARE Ctr, Los Angeles, California
  - Univ of California, San Diego, San Diego, California
  - University of California San Francisco, San Francisco, California
  - San Mateo County AIDS Program, Stanford, California
  - Stanford Univ, Stanford, California
  - Willow Clinic, Stanford, California
  - Univ of Colorado Health Sciences Ctr, Denver, Denver, Colorado
  - Howard Univ Hosp, Washington D.C., District of Columbia
  - North Broward Hosp District, Fort Lauderdale, Florida
  - Univ of Florida Health Science Ctr / Pediatrics, Jacksonville, Florida
  - Univ of Miami School of Medicine, Miami, Florida
  - Univ of Miami / Jackson Memorial Hosp, Miami, Florida
  - Univ of Miami (Pediatric), Miami, Florida
  - Emory Univ, Atlanta, Georgia
  - Univ of Hawaii, Honolulu, Hawaii
  - Mt Sinai Hosp Med Ctr / Dept of Pediatrics, Chicago, Illinois
  - Northwestern Univ Med School, Chicago, Illinois
  - The CORE Ctr, Chicago, Illinois
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Methodist Hosp of Indiana / Life Care Clinic, Indianapolis, Indiana
  - Wishard Hosp, Indianapolis, Indiana
  - Univ of Maryland (Pediatric), Baltimore, Maryland
  - Univ of Maryland, Institute of Human Virology, Baltimore, Maryland
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Boston Med Ctr (Harvard), Boston, Massachusetts
  - Boston Med Ctr (Pediatric), Boston, Massachusetts
  - Beth Israel Deaconess - West Campus, Boston, Massachusetts
  - Brigham and Women's Hosp, Boston, Massachusetts
  - Beth Israel Med Ctr, New York, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Columbia Presbyterian Med Ctr, New York, New York
  - Community Health Network, Rochester, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - State Univ of New York at Stony Brook, Stony Brook, New York
  - Montefiore Med Ctr Adolescent AIDS Program, The Bronx, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Duke Univ Med Ctr, Durham, North Carolina
  - Case Western Reserve Univ, Cleveland, Ohio
  - MetroHealth Med Ctr, Cleveland, Ohio
  - Univ of Pittsburgh, Pittsburgh, Pennsylvania
  - Brown Univ / Miriam Hosp, Providence, Rhode Island
  - Brown Univ / The Miriam Hosp, Providence, Rhode Island
  - Miriam Hosp / Brown Univ, Providence, Rhode Island
  - Julio Arroyo, West Columbia, South Carolina
  - University of Washington (Seattle), Seattle, Washington
- Puerto Rico (2):
  - Univ of Puerto Rico / Univ Children's Hosp AIDS, San Juan
  - San Juan City Hosp, San Juan